CLINICAL TRIAL: NCT05836350
Title: Targeting Branched-chain Amino Acid Oxidation to Improve Glycaemic Control in Patients With Type 2 Diabetes
Brief Title: Role of BCAA in Glucose Homeostasis
Acronym: NaPB2
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NaPB-2
Record Dates: First submitted 2023-04-07; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes
Keywords: type 2 Diabetes; branched-chain amino acid metabolism; glucose homeostasis; sodium-phenylbutyrate; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Clinical randomized controlled trial (RCT) with a double-blinded, placebo-controlled, cross-over design, including a wash-out period of 12 weeks. The trial will contain 2 treatment arms, with each a duration of 12 weeks.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4.8 g/m^2/day NaPB (Active Comparator): 12-week oral administration of 4.8 g/m^2/day Sodium-phenylbutyrate (NaPB) (in the form of Pheburane)
  Interventions: Drug: 4.8 g/m^2/day NaPB
- 4.8 g/m^2/day Placebo (Placebo Comparator): 12-week oral administration of 4.8 g/m2/day identical placebo granules.
  Interventions: Drug: 4.8 g/m^2/day placebo

INTERVENTIONS:
Drug: 4.8 g/m^2/day NaPB — 12-week oral administration of 4.8 g/m^2/day NaPB (in the form of Pheburane) per day. Although depending on body surface area, ~21 g Pheburane needs to be administered spread over the day in 3 times taken with a meal.
  Other Names: Pheburane; NaPB
  Arms: 4.8 g/m^2/day NaPB
Drug: 4.8 g/m^2/day placebo — 12-week oral administration of 4.8 g/m^2/day NaPB (in the form of Pheburane) or placebo per day. Although depending on body surface area, ~21 g Pheburane needs to be administered spread over the day in 3 times taken with a meal.
  Other Names: Placebo
  Arms: 4.8 g/m^2/day Placebo

SUMMARY:
This clinical trial study aims to evaluate the effects of prolonged NaPB treatment in a maximum of 20 patients with T2D. The primary objective is:

to investigate if prolonged boosting of ing BCAA oxidation will substantially lower plasma glucose levels in patients with T2D.

Participants will undergo a Clinical randomized controlled trial (RCT) with a double-blinded, placebo-controlled, cross-over design, including a wash-out period of 12 weeks. The trial will contain 2 treatment arms, with each a duration of 12 weeks.

Participants will have a 12-week oral administration of 4.8 g/m2/day NaPB (in the form of Pheburane) or placebo per day. Although depending on body surface area, ~21 g Pheburane needs to be administered spread over the day 3 times taken with a meal.

DETAILED DESCRIPTION:
Several studies identified branched-chain amino acids (BCAA; leucine, isoleucine, and valine) to be substantially elevated in people with T2D, possibly caused by lower BCAA oxidation rates. Plasma BCAA levels are strongly associated with insulin resistance and other key metabolic disarrangements as seen in T2D, including mitochondrial function, liver fat content, and metabolic flexibility. We, recently, showed that stimulating BCAA oxidation for 2 weeks with sodium-phenylbutyrate (NaPB) treatment -a drug known to accelerate BCAA oxidation- decreased BCAA plasma levels in patients with T2D. This reduction in plasma BCAA levels was paralleled with a robust improvement in peripheral insulin sensitivity and muscle mitochondrial oxidative capacity. Interestingly, a strong tendency was found for lower fasting glucose levels, an indication of better glucose control. These findings form lead to further evaluating this treatment strategy to improve glucose homeostasis and lower hyperglycaemic conditions in patients with T2D. So far, this strategy has been tested only in several rodent models reporting promising, beneficial outcomes on glucose homeostasis and heart function.

The aim of the present study is to evaluate the effects of prolonged treatment: patients with T2D will undergo a 12-week NaPB intervention with the aim of substantially lower fasting plasma glucose levels. The outcomes of this project evaluate a novel strategy to treat patients with T2D.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are able to provide signed and dated written informed consent prior to any study specific procedures
2. Women are post-menopausal (defined as at least 1 year post cessation of menses) and aged ≥ 45 and ≤ 76 years. Males are aged ≥ 40 years and ≤ 76 years
3. Patients should have suitable veins for cannulation or repeated venipuncture
4. Caucasians
5. BMI: 25-38 kg/m2
6. Diagnosed with T2D at least 1.5 years before the start of the study
7. Relatively well-controlled T2D: HbA1c < 8.5%
8. Oral glucose lowering medication: metformin only or in combination with sulfonylurea agents and/or on stable dose of a DPPIV inhibitor treatment for at least the last 3 months
9. No signs of active diabetes-related co-morbidities like active cardiovascular diseases, active diabetic foot, polyneuropathy or retinopathy
10. No signs of active liver or kidney malfunction

Exclusion Criteria:

1. Previous enrolment in a clinical study with an investigational product during the last 3 months or as judged by the Investigator
2. Participate in physical activity more than 3 times a week
3. Unstable body weight (weight gain or loss > 5 kg in the last three months)
4. Insulin dependent T2D
5. Patients with congestive heart failure and and/or severe renal and or liver insufficiency or known sodium retention with oedema
6. Patients using Probalan (probenecid), Haldol (haloperidol), Depakene (valproate) or medical products containing corticosteroids
7. Men: Hb <8.4 mmol/L, Women: Hb <7.8 mmol/l
8. Any contra-indication MRI scanning. These contra-indications include patients with e.g. the following:

   * Central nervous system aneurysm clip
   * Implanted neural stimulator
   * Implanted cardiac pacemaker of defibrillator
   * Cochlear implant
   * Metal containing corpora aliena in the eye or brains

Ages: 40 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
fasting plasma glucose levels | at week 12 of each intervention period
  Glucose levels will be measured after an overnight fast expressed in mmol/l.

SECONDARY OUTCOMES:
whole-body insulin sensitivity | at week 6 and week 12 of each intervention period
  glucose clearance in ml/kg determined during an OGTT at 6 weeks glucose disposal rate (delta Rd) in umol/kg/min measured with the clamp at 12 weeks
muscle mitochondrial function | at week 6 and week 12 of each intervention period
  O2-flux will be measured with high-resolution respirometry
whole-body metabolic flexibility | at week 12 of each intervention period
  insulin-stimulated change in respiratory exchange ratio will be determined with use of indirect calorimetry during the clamp
energy status of the heart | at week 12 of each arm
  PCr/ATP-ratio will be determined with phosphorus magnetic resonance spectroscopy
cardiac function: ejection fraction | at week 12 of each arm
  The cardiac function will be measured via ejection fraction (microL) with the use of cine-MRI
cardiac function: left atrial maximum volume | at week 12 of each arm
  The cardiac function will be measured via diastolic cardiac function with the use of ultrasound (transthoracic echocardiography) with the following parameter: Left atrial maximum volume (ml)
cardiac function: peak A-wave velocity (cm/sec) | at week 12 of each arm
  The cardiac function will be measured via diastolic cardiac function with the use of ultrasound (transthoracic echocardiography) with the following parameter: Peak A-wave velocity (cm/sec)
cardiac function: pulsed wave TDI velocity (cm/sec) at lateral and septal basal regions | at week 12 of each arm
  The cardiac function will be measured via diastolic cardiac function with the use of ultrasound (transthoracic echocardiography) with the following parameter: Pulsed wave TDI velocity (cm/sec) at lateral and septal basal regions
cardiac function: peak E-wave velocity | at week 12 of each arm
  The cardiac function will be measured via diastolic cardiac function with the use of of ultrasound (transthoracic echocardiography) will be assessed with the following parameters: Peak E-wave velocity (cm/sec)
cardiac function: tricuspid regurgitation systolic jet velocity | at week 12 of each arm
  The cardiac function will be measured via diastolic cardiac function with the use of ultrasound (transthoracic echocardiography) with the following parameter: Tricuspid regurgitation systolic jet velocity (m/sec)

IPD SHARING:
Plan to Share IPD: No